CLINICAL TRIAL: NCT00471055
Title: Efficacy Study on Symptomatic Control of Patient With Knee Osteoarthritis Between 0.0125% of Capsaicin to Placebo
Acronym: OAknee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Bangkok Laboratories and Cosmetics (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Khonkaen-ortho 1
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis, Knee Joint; Capsicum
Keywords: osteoarthritis; knee; capsaicin gel; capsicum
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Capsaicin and placebo controlled,Cross-over design study
  Interventions: Drug: 0.0125% Capsaicin gel "CAPSIKA gel"
- B (Placebo Comparator): Capsaicin and placebo controlled,Cross-over design study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 0.0125% Capsaicin gel "CAPSIKA gel"
  Arms: A
Drug: Placebo — Placebo
  Arms: B

SUMMARY:
The purpose of this study is to determine whether capsaicin gel is effective in treating mild to moderate degrees of osteoarthritis of the knee in the elderly patient compared with placebo gel.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis in the population. It is characterized pathologically by both focal loss of articular cartilage and marginal and central new bone formation. OA of knee, the principal large joint to be affected, results in disabling knee symptoms in an estimated 10% of people older than 55 years, a quarter of whom are severely disabled. The risk of disability attributable to knee OA alone is as great as that due to cardiac disease and greater than that due to any other medical disorder in the elderly. A recent World Health Organization report on the global burden of disease indicates that knee OA is likely to become the fourth most important global cause of disability in women and the eighth most important in men. Knee OA is associated with symptoms of pain and functional disability. Physical disability arising from pain and loss of functional capacity reduces quality of life and increases the risk of further morbidity and mortality. Current treatments aim at alleviating these symptoms of mild to moderate OA by several different methods: non-pharmacological treatment (for example education, exercise, lifestyle changes) or pharmacological treatments(for example paracetamol, NSAIDs and Capsaicin gel topical treatments). Current evidence to support the various treatments in current use, however, is very variable. Capsaicin, the active principle of hot chili pepper, is thought to selectively stimulate unmyelinated C fibre afferent neurons and cause the release of substance P. Prolonged application of capsaicin reversibly depletes stores of substance P, and possibly other neurotransmitters, from sensory nerve endings. This reduces or abolishes the transmission of painful stimuli from the peripheral nerve fibres to the higher centres.There were many study on Capsaicin gel to confirm the effectiveness of capsaicin gel in many dosages. However, there has been no efficacy study on the capsaicin 0.0125% of the Thai produce "Capsika gel " before, therefore, this study is proposed.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment in the study must meet all of the following criteria:

1. Subjects who are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
2. Ambulatory nom pregnant females and males 40-<80 years of age.
3. Subjects who withdraw pain medication or nutritional supplements for symptom relief for knee OA for a total of at least 15 days before screening visit 0.
4. Pain at or below 80 mm on a 100 mm VAS in the index knee.
5. A documented diagnosis of OA of the knee, or meeting American College of Rheumatology (ACR) clinical criteria for classification of idiopathic (primary) OA for at least 6 months prior to screening. If OA is presented in both knees the investigator will identify which knee will be X-rayed for study entry, with preference for the knee with more severe pain (<80mm VAS).
6. Has documented radiographic evidence of OA of the knee from the screening Visit radiograph of grade 2 or 3 according to Kellgren and Lawrence Radiographic Grading.
7. Subjects with baseline minimum joint space width in the medial compartment of the index knee of > 1.5 mm at Baseline, measured from radiographs using the MTP view.
8. Subjects with baseline minimum joint space width in the lateral compartment of the index knee of > 2.5 mm at Baseline, measured from radiographs using the MTP view.
9. Subject is able to understand and complete pain/function, global arthritis evaluation, and health outcome assessment.

Exclusion Criteria:

Subjects with any of the following criteria must not be enrolled in the study:

1. Subjects with history of hypersensitivity to capsaicin.
2. Subjects with skin lesion at the index knee.
3. A history of lower extremity surgery within 6 months prior to screening V0.
4. Significant prior injury to the index knee within 12 months prior to screening V0.
5. Disease of the spine or other lower extremity joints of sufficient degree to affect the index knee.
6. Treatment with other drugs potentially affecting bone or cartilage metabolism as described below:

   * chronic systematic corticosteroids
   * hyaluronan injection into the index knee with in the previous 6 months.
   * Diacerin treatment within the last 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
VAS and WOMAC | 8 months
VAS and WOMAC | 8-month study

CONTACTS AND LOCATIONS:
Overall Officials: weerachai Kosuwon, M.D, Principal Investigator — Department of Orthopedics, Faculty of Medicine, Khon kaen University
Locations (1):
- Weerachai Kosuwon, Khon Kaen University, Changwat Khon Kaen, Thailand